CLINICAL TRIAL: NCT01964144
Title: An Open-label, Multicenter, Phase II Study of Dovitinib in Advanced Thyroid Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2012-0405
Record Dates: First submitted 2013-10-09; First posted 2013-10-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Thyroid Cancer
Keywords: thyroid cancer, dovitinib
MeSH Terms: conditions — Thyroid Neoplasms | interventions — 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dovitinib arm (Experimental)
  Interventions: Drug: Dovitinib

INTERVENTIONS:
Drug: Dovitinib — Dovitinib 500mg (5 capsules x 100 mg/day) for 5 consecutive days and 2 days rest

SUMMARY:
There has been no effective treatment for advanced thyroid cancer that is not amenable to surgery and that does not concentrate iodine. Response rates with chemotherapy have been so low that best supportive care has been the standard of care for most patients. In recent phase I and phase II clinical studies, dovitinib has shown activity as a single agent in solid tumors. Therefore, we will conduct a phase II, single-arm trial to determine the efficacy of dovitinib in radioactive iodine-refractory recurrent or metastatic thyroid cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of thyroid cancer (papillary, follicular/Hürthle cell variant, medullary)
* Patients with metastatic or unresectable thyroid cancer for which curative measures (surgical resection, external-beam radiation therapy, or radioactive iodine) were no longer effective
* Documented evidence of disease progression (based on radiographic imaging), according to Response Evaluation Criteria in Solid Tumors (RECIST) criteria, within 6 months before entry into the study for papillary follicular/Hürthle cell variant
* Prior therapy with surgery, 131I treatment, chemotherapy, radiotherapy will be allowed, but not within 3 weeks of treatment.
* Patients who received a prior biologic treatment (kinase inhibitor, vaccine or antibody-based therapy), except prior VEGFR/FGFR inhibitor therapy, can be allowed after 3 weeks of treatment.
* Patients must have at least one measurable lesion, which has not been externally irradiated, as defined by RECIST criteria version 1.1
* Age : 20-90
* Performance status of Eastern Cooperative Oncology Group 0 to 2
* Life expectancy > 3 months
* Adequate bone marrow function: ANC≥1,500/uL, hemoglobin≥9.0 g/dL (can be corrected by transfusion) and platelet≥100,000/uL
* Adequate renal function (creatinine<1.5 mg/dL)
* Adequate liver function (total bilirubin <1.5 x ULN, trans-aminase <3 x ULN)
* Adequate blood glucose and lipid level (at fasting cholesterol < 2xUNL, triglyceride < 2xUNL, HbA1c < 9%)
* Patient compliance and geographic proximity that allow adequate follow up

Exclusion Criteria:

* Patients with CNS metastases
* Patients with another primary malignancy within 3 years prior to starting study drug, with the exception of adequately treated in-situ carcinoma of the uterine cervix, or skin cancer (such as basal cell carcinoma, squamous cell carcinoma, or non-melanomatous skin cancer)
* Patients who have received the last administration of an anticancer therapy including chemotherapy, immunotherapy, hormonal therapy and monoclonal antibodies (but excluding nitrosurea, mitomycin-C, targeted therapy and radiation) ≤ 4 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received the last administration of nitrosurea or mitomycin-C ≤ 6 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have received targeted therapy (e.g. sunitinib, sorafenib, pazopanib) ≤ 2 weeks prior to starting study drug, or who have not recovered from the side effects of such therapy
* Patients who have had radiotherapy ≤ 4 weeks prior to starting study drug, or ≤ 2 weeks prior to starting study drug in the case of localized radiotherapy (e.g. for analgesic purpose or for lytic lesions at risk of fracture), or who have not recovered from radiotherapy toxicities
* Pregnant or breast-feeding women
* Fertile males not willing to use contraception, as stated above
* Patients unwilling or unable to comply with the protocol

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 1 month after treatment
  Lesions measurements are performed by CT or MRI scan, evaluation by RECIST criteria v1.1

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Yonsei Cancer Center, Yonsei University College of Medicine, Seoul, South Korea